CLINICAL TRIAL: NCT04113018
Title: LCI-HEM-MYE-KRdD-001: Phase II Study of Daratumumab Combined With Carfilzomib, Lenalidomide and Dexamethasone in Newly Diagnosed Multiple Myeloma
Brief Title: Study of Daratumumab Combined With Carfilzomib, Lenalidomide and Dexamethasone for Newly Diagnosed Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Amgen (Industry); Celgene (Industry); Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00081541; 00037709 (Other: Advarra IRB); LCI-HEM-MYE-KRDD-001 (Other: Atrium Health)
Record Dates: First submitted 2019-09-27; First posted 2019-10-02 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Lenalidomide; Dexamethasone; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KRd-Daratumumab (Experimental): Induction: Carfilzomib, lenalidomide, dexamethasone (KRd) + Daratumumab
  Interventions: Drug: Carfilzomib, lenalidomide, dexamethasone (KRd) + Daratumumab

INTERVENTIONS:
Drug: Carfilzomib, lenalidomide, dexamethasone (KRd) + Daratumumab — Experimental

SUMMARY:
This study is being done because, despite major advances in therapy, MM is still considered an incurable disease. The purpose of this study is to determine the efficacy (how well it works) of the study treatment that combines the following drugs: daratumumab, carfilzomib, lenalidomide, dexamethasone in subjects who have a recent diagnosis of multiple myeloma (MM). Normal plasma (blood) cells are found in the bone marrow and are an important part of the immune system. MM is a cancer formed by malignant (cancerous) plasma cells. Daratumumab, one of the study drugs, is a man-made protein that works with your immune system by attaching itself to the cancerous cells. Once daratumumab attaches itself to these cells, it gets your body's immune system to attack and destroy the MM cells. Daratumumab has shown to be effective in subjects with MM when combined with medicines like bortezomib, or lenalidomide + dexamethasone.

DETAILED DESCRIPTION:
This single arm, two-stage, open-label Phase II study is designed with the primary objective of evaluating the efficacy of induction therapy comprised of 8 cycles of carfilzomib, lenalidomide, dexamethasone and daratumumab (KRd+daratumumab) in terms of complete response or better (CR) in subjects with NDMM, and comparing to relevant historical controls. Post induction, all subjects will undergo disease evaluation, including assessment of minimal residual disease (MRD). Post-induction disease evaluation will be followed by an MRD-based treatment algorithm. This trial will allow us to gather preliminary data on use of MRD status to direct post-induction therapy.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

1. Written informed consent and HIPAA authorization for release of personal health information signed by the subject or his/her legally authorized representative. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2 (see Appendix A, Section 18.1) within 28 days prior to day 1 of treatment.
4. Confirmation of newly diagnosed multiple myeloma (NDMM) as per the IMWG 2014 criteria (see Appendix D, Section 18.4). Newly diagnosed MM patients who may have deferred transplant are also allowed.
5. Measurable disease present at baseline assessments. Baseline disease assessments are defined as disease assessments collected within 28 days of initiation of the first pre-study induction cycle (subjects who received prior therapy) or within 28 days prior to day 1 of study treatment (subjects with no prior therapy). Measurable disease is defined as:

   1. Serum M-protein ≥ 1 g/dL (> 0.5 g/dL for IgA or IgM) OR
   2. Urine M-protein ≥ 200 mg/24 h OR
   3. Involved free light chain (FLC) level ≥ 10 mg/dL provided serum FLC ratio is abnormal
6. No more than one prior cycle of systemic therapy (completed within 6 weeks of consent) for MM (to accommodate subjects who needed emergent therapy at diagnosis); any prior radiotherapy must be completed at least 14 days prior to day 1 of treatment. Subject must have recovered from treatment-induced toxicities to ≤ grade 1 or baseline.
7. Demonstrate adequate organ function within 1 week of day 1 of treatment as defined in the table below:

   Hematological:
   * White Blood Cell (WBC) : ≥ 2,000/mm3
   * Absolute Neutrophil Count (ANC) : ≥ 1,000/mm3 without growth factors within 1 week of day 1 of treatment
   * Hemoglobin (Hgb) : ≥ 8 g/dL
   * Platelet count : ≥ 70,000/mm3 if bone marrow plasmacytosis of <50%; otherwise ≥ 50,000/mm3

   Renal:

   Serum creatinine with Creatinine clearance : ≤ 1.5 × upper limit of normal (ULN) with creatinine clearance

   ≥ 30 mL/min as measured by a 24-hour urine collection or estimated by the Cockcroft - Gault formula ( See formula in Appendix B, Section 18.2 )

   Hepatic:
   * Bilirubin : ≤ 2 × ULN; < 3.0 for subjects with Gilbert's Syndrome
   * Aspartate aminotransferase (AST) : ≤ 2.5× ULN
   * Alanine aminotransferase (ALT) : ≤ 2.5 × ULN
8. Adequate cardiac function as defined by ≥ 45% Left Ventricular Ejection Fraction (LVEF) by ECHO or MUGA within 28 days prior to day 1 of treatment.
9. Females of childbearing potential (FCBP) must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to day 1 of treatment, and be willing to undergo serial serum or urine pregnancy testing. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are postmenopausal (at least 12 consecutive months with no menses without an alternative medical cause).
10. FCBP must be willing to use a highly effective contraceptive method (i.e., achieves a failure rate of <1% per year when used consistently and correctly) plus a second contraceptive method (considered acceptable [failure rate of >1% per year] or highly effective) from the time of informed consent until 3 months after the last protocol prescribed therapy (which also includes FCBP on carfilzomib) has been discontinued. NOTE: estrogens may further increase the risk of thrombosis (beyond that associated with lenalidomide) and their use should be based on a benefit-risk decision. For the highly effective contraceptive method, a method with low user dependency is preferable but not required (see tables, adapted from: http://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf)

    Highly Effective Birth Control Methods:
    * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation

      * oral
      * intravaginal
      * transdermal
    * progestogen-only hormonal contraception associated with inhibition of ovulation

      * oral
      * injectable
      * implantable (Contraception method considered to have low user dependency)
    * intrauterine devide (IUD) (Contraception method considered to have low user dependency)
    * intrauterine hormone-releasing system (IUS) (Contraception method considered to have low user dependency)
    * vasectomised partner (Contraception method considered to have low user dependency) Vasectomised partner is a highly effective birth control method provided that partner is the sole sexual partner of the FCBP trial participant
    * sexual abstinence (Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments)

    Acceptable Birth Control Methods:
    * Progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action
    * Male or female condom with or without spermicide (A combination of male condom with either cap, diaphragm or sponge with spermicide (double barrier methods) are also considered acceptable, but not highly effective, birth control methods.
11. Male subjects (even those who have had a vasectomy) who are sexually active with a FCBP must be willing to use latex or synthetic condoms from initiation of study treatment until 3 months after the last protocol prescribed therapy has been discontinued. They must also refrain from donating sperm for at least 90 days after the last dose of carfilzomib and at least 90 days from the last dose of daratumumab. The FCBP partner should also consider contraception recommendations (see inclusion #10).
12. As determined by the enrolling physician, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

1. Any infection requiring systemic therapy (i.e. involving IV antibiotics) (NOTE: at discretion of investigator, subjects with uncomplicated urinary tract infections may be eligible).
2. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study, and any female subject must agree not to donate eggs during the study and for 3 months after the last protocol prescribed therapy has been discontinued).
3. Has a known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, carcinoma of the prostate with a current PSA value of <0.5 ng/mL or other cancer for which the subject has completed treatment, been disease-free for at least five years, and is considered by Sponsor-Investigator to be at <30% risk of relapse, or on hormonal therapy for a history of either prostate cancer or breast cancer, provided that there has been no evidence of disease progression during the previous three years.
4. Non-secretory MM.
5. Active involvement of the central nervous system by MM.
6. Prior cardiovascular cerebrovascular accident with persistent neurological deficit.
7. Has chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal. FEV1 is required for subjects suspected of having chronic obstructive pulmonary disease and are not eligible if FEV1 is < 50% of predicted normal.
8. Has had moderate or severe persistent asthma within the past 2 years from enrollment and/or has currently uncontrolled asthma of any classification. Note that participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate.
9. POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
10. Had major surgery within 2 weeks prior to day 1 of treatment.
11. Exposure to any investigational drug (including investigational vaccine) or invasive investigational medical device within 4 weeks or 5 pharmacokinetic half-lives prior to day 1 of treatment, whichever is longer.
12. Uncontrolled clinically significant illness including, but not limited to, uncontrolled hypertension (as per the most updated Joint National Committee for the Management of Hypertension definitions), symptomatic congestive heart failure (as per New York Heart Association [NYHA] class III or IV [see Appendix C, Section 18.3], uncontrolled angina pectoris, myocardial infarction within the past 6 months from consent, known or suspected amyloidosis, uncontrolled cardiac arrhythmia, psychiatric illness/social situations that would limit compliance with study requirements as determined by the investigator, or any other condition (including laboratory abnormalities) that would, in the opinion of the investigator, place the subject at unacceptable risk if he/she were to participate in the study.
13. Known allergies, hypersensitivity or intolerance to monoclonal antibodies or human proteins, daratumumab +hyaluronidase or its excipients or known sensitivity to mammalian-derived products, carfilzomib or its excipients, lenalidomide or its excipients, or dexamethasone or its excipients.
14. Is seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (i.e. subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. Exception: subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of HBV vaccination do not need to be tested for HBV DNA by PCR.
15. Is known to be seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy). Subject is not required to have hepatitis C testing at screening.
16. Is known to be seropositive for human immunodeficiency virus.
17. Transplant ineligible subjects > 70 years old only: Defined frail, per IMWG criteria of 'frailty'. Frailty assessment does not need to be performed unless the subject is transplant ineligible and > 70 years old. "Frail" is defined as a frailty score of ≥ 2.
18. Prior or current exposure to daratumumab or other anti-CD-38 therapies.
19. Focal radiation therapy within 14 days prior to C1D1 with the exception of palliative radiotherapy for symptomatic management but not on measurable extramedullary plasmacytoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2027-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Bhutani, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

REFERENCES:
- [Derived] Bhutani M, Robinson M, Foureau D, Atrash S, Paul B, Guo F, Grayson JM, Ivanina-Foureau A, Pineda-Roman M, Varga C, Friend R, Ferreri CJ, Begic X, Norek S, Drennan T, Anderson MB, Symanowski JT, Voorhees PM, Usmani SZ. MRD-driven phase 2 study of daratumumab, carfilzomib, lenalidomide, and dexamethasone in newly diagnosed multiple myeloma. Blood Adv. 2025 Feb 11;9(3):507-519. doi: 10.1182/bloodadvances.2024014417. PMID 39576965

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | KRd-Daratumumab
Started | 39
Completed | 0
Not Completed | 39
Not completed — Death | 2
Not completed — Lost to Follow-up | 1
Not completed — Still On Study (on study treatment) | 24
Not completed — Still On Study (in follow up) | 12

BASELINE CHARACTERISTICS:
Arm/Group | KRd-Daratumumab
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 16
Age, Continuous [Median (Full Range); unit: years] | 62 [34 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response or Stringent Complete Response to Induction
Description: The primary endpoint is a binary variable determined for each subject indicating whether the subject achieved a complete response (CR) or stringent complete response (sCR) to induction treatment with KRd-Dara, as defined by the IMWG 2016 response criteria. Per IMWG 2016 criteria, CR is defined as negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow aspirates. sCR is defined as CR plus normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry.
Time Frame: From enrollment to best response determined at the end of induction (8 28-day cycles); the median length of induction was 32 weeks
Population: The response evaluable population is defined as all subjects who initiate treatment with daratumumab and who have measurable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | KRd-Daratumumab
Number analyzed (Participants) | 39
Participants | 21
Statistical Analysis 1: Comparison: KRd-Daratumumab; A minimax 2-stage design was used to test the hypothesis that the CR+ rate less than or equal to 50%. Twenty-three evaluable subjects were enrolled in the first stage, followed by an additional 16 subjects for a total of 39 subjects. This design provided 90% power to detect a difference of 20% under the alternative hypothesis, assuming a one-sided alpha=0.10 significance level. If at least 24 of 39 participants had achieved CR or better to induction, the null hypothesis would have been rejected; Test type: Superiority; p = 0.375, Fisher Exact; Response rate = 0.5385, 95% CI 2-sided [0.3718 to 0.6991] — Confidence interval estimated using the Clopper Pearson method

2. Secondary Outcome: Number of Participants With an Objective Response (OR)
Description: Objective response is determined for each subject as a binary variable indicating whether or not the subject achieved a best overall response of stringent complete response (sCR), complete response (CR) or partial response (PR) as determined by IMWG 2016 response criteria.
Time Frame: From enrollment to best response while on study treatment; subjects remained on treatment until disease progression or death or unacceptable toxicity; assessed for approximately 5 years
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the duration from enrollment to the study (treatment start date) to the date of death from any cause. Participants who are alive or lost to follow-up at the time of the analysis will be censored at the last known date they were alive.
Time Frame: From date of treatment start to date of death, or censored as described; assessed for approximately 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from treatment start date to first occurrence of either progressive disease (PD) or death. PD must be objectively determined per IMWG 2016 criteria, where progression date is date of last assessment that identified PD. If subject died without documented PD, progression date will be death date. For surviving subjects who do not have PD, PFS will be censored at the date of last disease assessment. For subjects who received subsequent anti-cancer therapy prior to documented PD, PFS will be censored at the date of last disease assessment prior to commencement of subsequent therapy. Subjects who have an initial PFS event immediately following 2 or more consecutive missed assessments will be censored at date of last assessment prior to missed assessments.
Time Frame: From date of treatment start to date of progression or death, or censored as described; assessed for approximately 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Time to Disease Progression (TTP)
Description: TTP is defined as the duration of time from treatment start date to first occurrence of either progressive disease (PD) or death related to disease progression. PD must be objectively determined per IMWG 2016 criteria, where progression date is date of last assessment that identified PD. If a subject died for causes related to disease progression then progression date will be date of death. If a subject died for causes other than disease progression, TTP will be censored at the date of other cause mortality. For surviving subjects who do not have PD, TTP will be censored at the date of last disease assessment. For subjects who received subsequent anti-cancer therapy prior to documented PD, TTP will be censored at the date of last disease assessment prior to commencement of subsequent therapy. Subjects who have an initial TTP event immediately following 2 or more consecutive missed assessments will be censored at date of last assessment prior to missed assessments.
Time Frame: From date of start of treatment to date of disease progression or death, or censored as described; assessed for approximately 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response (DoR) will be calculated for each subject achieving a PR or better and will be calculated from the time of the first assessment that identified response until disease progression or death. The censoring mechanism will be the same as described for PFS.
Time Frame: From date of first response to date of progression or death, or censored as described; assessed for approximately 5 years
Reporting Status: Not Posted

7. Secondary Outcome: Time to Next Treatment (TTNT)
Description: Time to next treatment (TTNT) will be calculated from the time of treatment start until the start of the first subsequent anti-cancer therapy after all protocol directed therapy is completed. For surviving subjects who do not receive subsequent therapy, TTNT will be censored at the last contact date. For subjects who die before beginning subsequent anti-cancer therapy, TTNT will be censored at the date of death.
Time Frame: From treatment start date to date of next treatment, or censored as described; assessed for approximately 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Number of Participants With Grade 3 or Higher Treatment-related Cardiovascular or Pulmonary-related Adverse Events During Induction
Description: A binary variable will be determined for each subject indicating whether or not the subject experienced at least one grade 3 or higher study treatment-related cardiovascular or pulmonary-related adverse event according to the NCI Common Terminology for Adverse Events version 4.03 during induction. Only select CTCAE terms will be considered for this safety outcome including heart failure, pneumonia, dyspnea, peripheral edema, or hypertension.
Time Frame: From enrollment to completion of induction; evaluated for approximately 32 weeks (8 28-day cycles).
Population: The evaluable population is defined as all subjects who initiate treatment with daratumumab.
Measure: Count of Participants; unit: Participants
Arm/Group | KRd-Daratumumab
Number analyzed (Participants) | 39
Participants | 2
Statistical Analysis 1: Comparison: KRd-Daratumumab; Test type: Other — Estimation only; Rate = 0.0513, 95% CI 2-sided [0.0063 to 0.1732] — Confidence interval estimated using the Clopper Pearson method

9. Other Pre Specified Outcome: Number of Participants With Grade 5 Adverse Events During Induction
Description: A binary variable will be determined for each participant indicating whether or not the subject died due to an adverse event during induction. This will include any grade 5 adverse event (according to NCI Common Terminology for Adverse Events version 4.03), regardless of causality
Time Frame: From enrollment to completion of induction; evaluated for approximately 32 weeks (8 28-day cycles).
Population: The evaluable population is defined as all subjects who initiate treatment with daratumumab.
Measure: Count of Participants; unit: Participants
Arm/Group | KRd-Daratumumab
Number analyzed (Participants) | 39
Participants | 1
Statistical Analysis 1: Comparison: KRd-Daratumumab; Test type: Other — Estimation only; Rate = 0.0256, 95% CI 2-sided [0.0006 to 0.1348] — Confidence interval estimated using the Clopper Pearson method

10. Other Pre Specified Outcome: Number of Participants With at Least One Serious Adverse Event
Description: A binary variable will be determined for each participant indicating whether or not the subject had at least one adverse event that was categorized as serious, regardless of causality. Serious is defined per the study protocol and includes events that the investigator deems serious and results in the following outcomes: death, life-threatening situation, persistent or significant disability/incapacity, requires or prolongs hospitalization, congenital anomaly/birth defect in the offspring of a study participant, suspected transmission of any infectious agent via medial product, or based upon medical judgement, may jeopardize the subject and may require medical or surgical intervention to prevent one of the afore listed outcomes from occurring.
Time Frame: From enrollment to 30 days following cessation of study treatment. Reasons for study treatment discontinuation include progression, toxicity, consent withdrawal, or investigator decision; assessed for approximately 5 years.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Number of Participants With at Least One Treatment Emergent Adverse Event
Description: A binary variable will be determined for each participant indicating whether or not the subject had at least one treatment-emergent adverse event, regardless of causality. Adverse events will be categorized per NCI Common Terminology for Adverse Events version 4.03. Treatment-emergent is defined per the study protocol and includes AEs that occur after treatment start that were not present at the time of treatment start or AEs that increase in severity after treatment start if the event was present at the time of treatment start.
Time Frame: as for outcome 10
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Number of Participants With at Least One Grade 3 or Higher Treatment Emergent Adverse Event
Description: A binary variable will be determined for each participant indicating whether or not the subject had at least one grade 3 or higher treatment-emergent adverse event, regardless of causality. Adverse events will be categorized per NCI Common Terminology for Adverse Events version 4.03. Treatment-emergent is defined per the study protocol and includes AEs that occur after treatment start that were not present at the time of treatment start or AEs that increase in severity after treatment start if the event was present at the time of treatment start.
Time Frame: as for outcome 10
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Number of Participants Who Discontinued Study Treatment Due to Adverse Events
Description: A binary variable will be determined for each participant indicating whether or not the subject discontinued study treatment due to adverse events.
Time Frame: as for outcome 10
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Daratumumab Administration - Number of Cycles Received
Description: Descriptive summary of daratumumab administration. Number of cycles of daratumumab received.
Time Frame: From enrollment to completion of induction; evaluated for approximately 32 weeks (8 28-day cycles).
Population: The evaluable population is defined as all subjects who initiate treatment with daratumumab
Measure: Median (Full Range); unit: count of cycles
Arm/Group | KRd-Daratumumab
Number analyzed (Participants) | 39
count of cycles | 7 [1 to 8]

15. Other Pre Specified Outcome: Daratumumab Administration - Number of Doses Received
Description: Descriptive summary of daratumumab administration. Number of doses of daratumumab received.
Time Frame: From enrollment to completion of induction; evaluated for approximately 32 weeks (8 28-day cycles).
Population: The evaluable population is defined as all subjects who initiate treatment with daratumumab
Measure: Median (Full Range); unit: count of doses
Arm/Group | KRd-Daratumumab
Number analyzed (Participants) | 39
count of doses | 17 [1 to 19]

ADVERSE EVENTS:
Time Frame: Baseline, during treatment, and through 30 days after study treatment is discontinued, an average of 27 months.
Arm/Group | KRd-Daratumumab
All-Cause Mortality (participants affected / at risk) | 2/39
Serious Adverse Events (participants affected / at risk) | 15/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KRd-Daratumumab (N=39)
Anemia (Blood and lymphatic system disorders) | 1
Heart failure (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Fever (General disorders and administration site conditions) | 4
Pain (General disorders and administration site conditions) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Sepsis (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 1 — infection blood
Infections and infestations - Other (Infections and infestations) | 1 — COVID-19
Lung infection (Infections and infestations) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 — Knee replacement surgery
Intracranial hemorrhage (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 — Pneumonia
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 — Community-acquired pneumonia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KRd-Daratumumab (N=39)
Anemia (Blood and lymphatic system disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 4
Palpitations (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Cardiac disorders - Other (Cardiac disorders) | 1 — premature atrial complexes
Cardiac disorders - Other (Cardiac disorders) | 1 — intermittent chest tightness
Sinus tachycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Hearing impaired (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Endocrine disorders - Other (Endocrine disorders) | 1 — thyroid nodule
Blurred vision (Eye disorders) | 7
Conjunctivitis (Eye disorders) | 3
Cataract (Eye disorders) | 1
Eye disorders - Other (Eye disorders) | 1 — blepharitis
Eye disorders - Other (Eye disorders) | 1 — blepharoconjuncivits
Eye disorders - Other (Eye disorders) | 1 — burning eyes
Eye disorders - Other (Eye disorders) | 1 — plugged tear duct
Eye disorders - Other (Eye disorders) | 1 — posterior virteous detachment
Eye disorders - Other (Eye disorders) | 1 — red tear ducts swollen
Eye disorders - Other (Eye disorders) | 1 — Right eye stye on upper eyelid
Eye disorders - Other (Eye disorders) | 1 — Sty Left Eyelid
Floaters (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Watering eyes (Eye disorders) | 1
Diarrhea (Gastrointestinal disorders) | 25
Constipation (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 10
Abdominal pain (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Bloating (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Stomach pain (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Fecal incontinence (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 — abdominal ache
Ileus (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 — Abdominal bloating
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 — diverticulitis
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 — fecal frequency
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 — gastroenteritis
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 — stomach upset
Fatigue (General disorders and administration site conditions) | 14
Edema limbs (General disorders and administration site conditions) | 9
Chills (General disorders and administration site conditions) | 6
Fever (General disorders and administration site conditions) | 5
Infusion related reaction (General disorders and administration site conditions) | 5
Pain (General disorders and administration site conditions) | 4
Localized edema (General disorders and administration site conditions) | 3
Non-cardiac chest pain (General disorders and administration site conditions) | 2
Flu like symptoms (General disorders and administration site conditions) | 1
General disorders and administration site conditions - Other (General disorders and administration site conditions) | 1 — General pain
Cholecystitis (Hepatobiliary disorders) | 1
Immune system disorders - Other (Immune system disorders) | 1 — low immunoglobulin G
Upper respiratory infection (Infections and infestations) | 13
Infections and infestations - Other (Infections and infestations) | 11 — COVID-19
Urinary tract infection (Infections and infestations) | 4
Conjunctivitis infective (Infections and infestations) | 2
Gum infection (Infections and infestations) | 2
Lung infection (Infections and infestations) | 2
Nail infection (Infections and infestations) | 2
Skin infection (Infections and infestations) | 2
Enterocolitis infectious (Infections and infestations) | 1
Hepatitis viral (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 1 — bacteremia
Infections and infestations - Other (Infections and infestations) | 1 — Incision
Infections and infestations - Other (Infections and infestations) | 1 — shingles
Papulopustular rash (Infections and infestations) | 1
Penile infection (Infections and infestations) | 1
Phlebitis infective (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 8
Bruising (Injury, poisoning and procedural complications) | 3
Fracture (Injury, poisoning and procedural complications) | 2
Spinal fracture (Injury, poisoning and procedural complications) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 — Dog bite
Vascular access complication (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 14
Creatinine increased (Investigations) | 7
Blood bilirubin increased (Investigations) | 5
Platelet count decreased (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Investigations - Other (Investigations) | 1 — cT1C adenocarcinoma of the prostate
Investigations - Other (Investigations) | 1 — Elevated PSA
Investigations - Other (Investigations) | 1 — hip pain- right hip
Investigations - Other (Investigations) | 1 — Vitamin B12 deficiency
Weight gain (Investigations) | 1
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 11
Hypokalemia (Metabolism and nutrition disorders) | 10
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Hyperglycemia (Metabolism and nutrition disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 4
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 3 — Decreased Vitamin D Level
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 — Vitamin B12 deficiency
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 — muscle spasm
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 — intermittent muscle cramps
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 — hand cramping
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 — Right Foot Swelling
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 — Planned knee surgery
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 — Left hip pain
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 — Jaw Pain
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 — gout
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 — Cervical Spine Stenosis
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 — Bilateral hip stiffness
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — basal cell carcinoma
Peripheral sensory neuropathy (Nervous system disorders) | 9
Headache (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 6
Tremor (Nervous system disorders) | 6
Syncope (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 4
Paresthesia (Nervous system disorders) | 4
Presyncope (Nervous system disorders) | 3
Spasticity (Nervous system disorders) | 3
Lethargy (Nervous system disorders) | 2
Concentration impairment (Nervous system disorders) | 1
Extrapyramidal disorder (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Vasovagal reaction (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 8
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Urinary frequency (Renal and urinary disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 — BPH
Vaginal dryness (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — cat scratch to eye
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — contact dermatitis
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — erythema rash
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — laceration
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — Lower extremity rash
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — psoriasis
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — skin erythema
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — squamous cell carcinoma
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — wound on right shoulder
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 — wisdom teeth removal
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 6
Thromboembolic event (Vascular disorders) | 3
Hot flashes (Vascular disorders) | 2
Phlebitis (Vascular disorders) | 2
Superficial thrombophlebitis (Vascular disorders) | 2
Vascular disorders - Other (Vascular disorders) | 1 — bilateral deep vein thrombosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT04113018/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT04113018/ICF_000.pdf